CLINICAL TRIAL: NCT01818921
Title: Randomized, Double-Blind, Placebo Controlled, Parallel Dose Ranging Phase 2a Trial of ZGN-440 (Subcutaneous Beloranib in Suspension), A Novel Methionine Aminopeptidase 2 Inhibitor, in Over-weight and Obese Subjects With Prader-Willi Syndrome to Evaluate Weight Reduction, Food-related Behavior, Safety, and Pharmacokinetics Over 4 Weeks Followed by Optional 4-Week Open-Label Extension
Brief Title: An Efficacy, Safety, and Pharmacokinetics Study of Beloranib in Obese Subjects With Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zafgen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAF-211
Record Dates: First submitted 2013-03-21; First posted 2013-03-27 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2016-07

CONDITIONS: Obesity; Over-weight; Prader-Willi Syndrome
Keywords: Beloranib; ZGN-440; ZGN-440 for injectable suspension; ZGN-433
MeSH Terms: conditions — Obesity; Prader-Willi Syndrome | interventions — CKD732

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZGN-440 sterile diluent (Placebo Comparator): Subjects will receive placebo twice weekly subcutaneous injections for up to 6 weeks.
  Interventions: Drug: ZGN-440 sterile diluent
- 1.2 mg ZGN-440 for injectable suspension (Experimental): Subjects will receive ZGN-440 for injectable suspension (beloranib) twice weekly subcutaneous injections for up to 8 weeks.
  Interventions: Drug: 1.2 mg ZGN-440 for injectable suspension
- 1.8 mg ZGN-440 for injectable suspension (Experimental): Subjects will receive ZGN-440 for injectable suspension (beloranib) twice weekly subcutaneous injections for up to 8 weeks.
  Interventions: Drug: 1.8 mg ZGN-440 for injectable suspension

INTERVENTIONS:
Drug: ZGN-440 sterile diluent — ZGN-440 sterile diluent/placebo
  Other Names: Placebo
  Arms: ZGN-440 sterile diluent
Drug: 1.2 mg ZGN-440 for injectable suspension — 1.2 mg beloranib
  Other Names: ZGN-440 for injectable suspension; ZGN-440; ZGN-433; Beloranib
  Arms: 1.2 mg ZGN-440 for injectable suspension
Drug: 1.8 mg ZGN-440 for injectable suspension — 1.8 mg beloranib
  Other Names: ZGN-440 for injectable suspension; ZGN-440; ZGN-433; Beloranib
  Arms: 1.8 mg ZGN-440 for injectable suspension

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics for certain doses of beloranib in obese subjects with Prader-Willi Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Prader-Willi Syndrome due to chromosome 15 micro-deletion, maternal uniparental disomy, or imprinting defect
* BMI ≥25 kg/m2
* Type 2 diabetes mellitus is allowed
* Subject must agree to stay at the group home or under supervision of the group home or site staff (i.e. no home visits) for the duration of the study
* Stable body weight during the past 3 months, except for during home visits

Exclusion Criteria:

* Use of weight loss agents in the past 3 months
* Type 1 diabetes mellitus
* Current or anticipated chronic use of narcotics or opiates

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Percent change in body weight from baseline to the end of the randomized dosing period. | 4 weeks

SECONDARY OUTCOMES:
Change in body weight (kg) from baseline to the end of the randomized dosing period | 4 weeks
Change in hyperphagia behavior, drive, and severity score (total score) from baseline to the end of the randomized dosing period using the PWS Hyperphagia Questionnaire | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Miller, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States